CLINICAL TRIAL: NCT02039648
Title: Proanthocyanidin- Enriched Extract From Rumex Acetosa L. as a Prophylactic Agent Against Intraoral Colonization With Porphyromonas Gingivalis
Brief Title: The Influence of Rumex Acetosa L on the Intraoral Colonization With Porphyromonas Gingivalis
Acronym: RPG-I
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NRW 300262502
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Periodontitis
Keywords: Periodontitis; Porphyromonas gingivalis; Rumex acetosa L.; Proanthocyanidins
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rumex acetosa L. extract (Active Comparator): Rumex acetosa L. extract mouthrinse, 10 ml, tid, 3 min, 7 days
  Interventions: Other: Rumex acetosa L. extract
- Placebo (Placebo Comparator): Placebo mouthrinse, 10 ml, tid, 3 min, 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Rumex acetosa L. extract
  Arms: Rumex acetosa L. extract
Other: Placebo
  Arms: Placebo

SUMMARY:
Periodontitis is a biofilm depended oral infection. It leads to inflammatory destruction of periodontal tissues and if left untreated to tooth loss. Porphyromonas gingivalis (P.g.) is one of the major pathogens associated with the onset and progression of periodontitis. Previous in vitro studies have shown that a proanthocyanidin-enriched extract from Rumex acetosa L. inhibits the adhesion of P.g. and acts in a cytoprotective manner. Since the the bacterial adhesion to oral mucosa cells is a pivotal step for the P.g. mediated tissue destruction, its inhibition may be helpful in preventing the colonization with P.g. or its eradication in P.g. infected patients. Therefore, the aim of this controlled, randomized and double blinded study was to analyze the effects of a Proanthocyanidin-enriched extract from Rumex acetosa L. on the intraoral colonization with Porphyromonas gingivalis in individuals harboring P.g. intramurally.

DETAILED DESCRIPTION:
During screening phase plaque samples of healthy individuals were tested via polymerase chain reaction for the prevalence of P.g..

At baseline those identified P.g. positive participants received a supragingival debridement (professional tooth cleaning) and were randomly assigned to the test- or control-group. Afterwards the study participants are instructed to rinse 3 times per day with 10 ml of either Rumex acetosa L. extract mouth rinse or the placebo mouth rinse for 7 days in addition to their oral hygiene procedures. Plaque samples were taken at different visits (screening, baseline, 2, 4, 7 and 14 days after baseline) and P.g. was identified and quantified by real-time polymerase chain reaction (qrt-PCR). Also the relative quantity of eight other oral pathogenic microorganisms (Aggregatibacter actinomycetemcomitans, Treponema denticola, Tannerella forsythia, Prevotella nigrescens, Prevotella intermedia, Eikenella corrodens, Streptococcus mutans and Candida albicans) and four commensal bacteria (Streptococcus sanguinis, Streptococcus mitis, Veillonella parvula and Actinomyces viscosus) was determined over the whole study period by qrt-PCR. Additionally clinical parameters, i.e. the Approximal Plaque Index (API) and the modified Sulcular Bleeding Index (SBI) were recorded at baseline, 7 and 14 days. For identifying any dysplastic changes and mutations as a potential reaction to the tested mouthwash solutions brushing biopsies of the oral mucosa were taken at baseline and day 7 and were histologically examined.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* periodontally healthy with Periodontal Screening Index ≤ 2

Exclusion Criteria:

* antibiotic therapy within the previous 6 months
* allergies against mouthrinse components
* pregnancy or lactation
* soft tissue lesions (e.g. lichen planus, leukoplakia)
* history of periodontal disease and/ or PSI ≥ 3 or more
* any topical or systemical medication, that potentially influence any immunological parameters
* any systemic disease or medical condition (e.g. diabetes or immunological disorders), that potentially influence the immune response or compromise the study results
* any systemic conditions, that require an antibiotic coverage for routine dental procedures (e.g. endocarditis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
change of the intraoral prevalence of Porphyromonas gingivalis | change from baseline to 2, 4, 7 and 14 days

SECONDARY OUTCOMES:
change of the Approximal Plaque Index | change from baseline to 7 and 14 days
change of the Sulcular Bleeding Index | change from baseline to 7 and 14 days
change of the cytopathological appearance of the mucosal tissue | change from baseline to 7 days

OTHER OUTCOMES:
change of the intraoral prevalence of Aggregatibacter actinomycetemcomitans | change from baseline to 2, 4,7, and 14 days
change of the intraoral prevalence of Treponema denticola | change from baseline to 2, 4, 7, and 14 days
change of the intraoral prevalence of Tannerella forsythia | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Prevotella intermedia | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Prevotella nigrescens | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Eikenella corrodens | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Streptococcus mutans | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Candida albicans | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Streptococcus sanguinis | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Streptococcus mitis | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Veillonella parvula | change from baseline to 2, 4, 7 and 14 days
change of the intraoral prevalence of Actinomyces viscosus | change from baseline to 2, 4, 7 and 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Beikler, Prof., Principal Investigator — Heinrich-Heine-University
Locations (1):
- Department od Operative Dentistry, Periodontics and Endodontics, Düsseldorf, Germany